CLINICAL TRIAL: NCT01084629
Title: The Role of the Fujinon Intelligent Chromo Endoscopy (FICE™) for the Detection of Dysplasia in Barrett's Esophagus and in Post Ablation Barrett's Esophagus
Brief Title: The Role of the Fujinon Intelligent Chromo Endoscopy (FICE™) in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenneth K. Wang, Kathy and Russ Van Cleve Professor of Gastroenterology Research, Mayo Clinic
Other Study IDs: 07-006981
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Surveillance
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surveillance Barrett's esophagus: Patients scheduled for endoscopic surveillance of Barrett's esophagus
- Barrett's esophagus post ablation: Patients scheduled for surveillance endoscopy who have undergone ablative therapies (PDT, RF ablation) for their Barrett's esophagus

SUMMARY:
The purpose of this study to assess post ablation, if there are areas of Barrett's mucosa post ablation and to assess the ability of the Fujinon FICE system to detect this, as compared to white light endoscopy. A subgroup will also be compared with laser confocal microscopy

ELIGIBILITY:
Inclusion Criteria:

* Visible Barrett's esophagus
* Scheduled for Surveillance Endoscopy
* Able to undergo endoscopy

Exclusion Criteria:

* Unable to undergo endoscopy
* Unable to stop blood thinning medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Barrett's esophagus
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
detection of dysplasic areas | during surveillance endoscopy
  Areas of residual mucosa will be scored for being present, absent or suspicious. The ability of both FICE and white light endoscopy to find areas will be graded on the number of areas found, and the size of the areas estimated at the time of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials